CLINICAL TRIAL: NCT02078661
Title: A Single Center, Randomized, Double-Masked, Placebo Controlled Study Evaluating the Safety and Efficacy of 0.25% PG101 and 1.0% PG101 in Subjects With Dry Eye Syndrome
Brief Title: Safety and Efficacy of PG101 for Dry Eye Syndrome
Acronym: PG101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-PG-EF001; 13-110-0002 (Other: Rhodes Pharmaceuticals L.P.)
Record Dates: First submitted 2013-12-20; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Dry Eye Syndrome
Keywords: Keratoconjunctivitis sicca; Dry eye
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PG101 0.25% (Active Comparator): Topical application of drug
  Interventions: Drug: PG101
- PG101 1.0% (Active Comparator): Topical application of drug
  Interventions: Drug: PG101
- Placebo (Placebo Comparator): Topical application of placebo
  Interventions: Drug: PG101

INTERVENTIONS:
Drug: PG101 — A topical gel containing either 1% or 0.25% PG101 active.
  Other Names: Topical gel; Topical gel suspension

SUMMARY:
To evaluate the safety and efficacy of 0.25% PG101 and 1.0% PG101 topical gel suspension compared to placebo when administered two times daily for 14 days in subjects diagnosed with dry eye syndrome

DETAILED DESCRIPTION:
The topical product PG101 is expected to be efficacious in treating the symptoms of dry eye such as discomfort, dryness, grittiness, burning, stinging, photophobia, lid friction, mucus discharge and hyper-tearing. Two concentrations (0.25% and 1.0%) are included in the study to determine if there is a dose response effect.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female of any race, at least 18 years of age
* Have provided verbal and written informed consent
* Be able and willing to follow instructions, including participation in all study assessments and visits
* Have a reported history of dry eye syndrome
* Have a history of use or desire to use eye drops for dry eye
* If a woman of childbearing potential, have a negative pregnancy test at Visit 1 and be using an adequate method of birth control throughout the study period
* Have a best corrected visual acuity of +0.70 logMAR or better in both eyes

Exclusion Criteria:

* Have any clinically significant eye findings that require therapeutic treatment or may interfere with study parameters
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g. follicular conjunctivitis) at Visit 1
* Be a woman who is pregnant, nursing or planning a pregnancy
* Have a known allergy and/or sensitivity to the test article or its components
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
At least one dry eye ocular symptom | Up to 2 weeks
  Dry eye ocular symptoms measured are: Ocular discomfort, dryness, grittiness, burning, stinging, photophobia, lid friction, mucus discharge and hyper-tearing.

SECONDARY OUTCOMES:
At least one dry eye ocular sign measure. | Up to 2 weeks
  Dry eye ocular signs measured are: Corneal and conjunctival staining, tear break up time, OPI 2.0, Schirmer tear test, quality of life, and conjunctival redness

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, M.D., Principal Investigator — Andover Eye
Locations (1):
- Andover Eye, Andover, Massachusetts, United States